CLINICAL TRIAL: NCT06087211
Title: Pain Relieving Potentials of Preoperative Combination of Single Dose Oral Duloxetine and Intravenous Magnesium Sulphate in Acute and Chronic Post Mastectomy Pain: A Randomized Controlled Trial
Brief Title: Pain Relieving Potentials of Combination of Oral Duloxetine and Intravenous Magnesium Sulphate in Post Mastectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Norma Osama Abdalla Zayed, Lecturer of Anesthesia, Surgical ICU and Pain Management, National Cancer Institute, Cairo University, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP2307-301-002
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Duloxetine; Magnesium Sulphate; Post-mastectomy Pain Syndrome
MeSH Terms: interventions — Magnesium Sulfate; Duloxetine Hydrochloride; Magnesium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DM group (Active Comparator): Patients received Duloxetine 30mg orally and an intravenous infusion of magnesium sulphate 50mg/kg mixed with 200 ml of normal saline.
  Interventions: Drug: Magnesium sulphate and Duloxetine
- D group (Active Comparator): Patients received Duloxetine 30mg orally and 200 ml of normal saline.
  Interventions: Drug: Duloxetine
- Control group (Placebo Comparator): Patients received a placebo capsule and an intravenous infusion of 200 mL of normal saline
  Interventions: Drug: Placebo and normal saline

INTERVENTIONS:
Drug: Magnesium sulphate and Duloxetine — Patients received Duloxetine 30mg orally and an intravenous infusion of magnesium sulphate 50mg/kg mixed with 200 ml of normal saline.
  Other Names: magnesium and cymbalta
  Arms: DM group
Drug: Duloxetine — Patients received Duloxetine 30mg orally and 200 ml of normal saline.
  Other Names: cymbalta
  Arms: D group
Drug: Placebo and normal saline — Patients received a placebo capsule and an intravenous infusion of 200 mL of normal saline.
  Other Names: placebo
  Arms: Control group

SUMMARY:
This study aims to evaluate the effect of combined duloxetine and IV Magnesium sulphate to decrease acute and chronic post mastectomy pain.

The study will be conducted in National Cancer Institute and all the participants will be enrolled from female patients scheduled for modified radical mastectomy under general anesthesia in National Cancer Institute, Cairo University.

DETAILED DESCRIPTION:
It has been reported recently that Duloxetine improved the quality of recovery in patients subjected to hysterectomy. In this context, mastectomy has a negative consequence starting from cancer diagnosis to the squeal of cancer-related treatments and it has been estimated that 20%-30% of patients with breast cancer suffer from depression and anxiety. Magnesium also antagonizes the release of inflammatory mediators such as histamine, serotonin, and cytokines in peripheral tissues.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old.
* American Society of Anesthesiologists (ASA) physical I-II
* Scheduled for modified radical mastectomy (MRM) under general anesthesia.

Exclusion Criteria:

* Liver or kidney disease
* Patient with previous chronic pain on opioids
* Patients on antidepressants and antipsychotics.
* Allergies to study drugs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female scheduled for modified radical mastectomy
Enrollment: 90 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic request | 48 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administared).

SECONDARY OUTCOMES:
Total morphine consumption | 48 hours postoperatively
  Postoperative analgesia is composed of PCA-morphine, set to deliver 2 mg boluses on-demand without background infusion with a lockout period of 10 min and regular intravenous paracetamol, one gram every 8 h.
Degree of pain | 48 hours postoperatively
  Each patient was instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at post-anesthesia care unit (PACU), 1, 2, 4, 6, 8, 12, 24, 36 and 48 h postoperatively.
Incidence of post-mastectomy pain syndrome | 12 weeks postoperatively
  Incidence of post-mastectomy pain syndrome was determined at 8- and 12-weeks post-mastectomy.
Degree of patient satisfaction | 48 hours postoperatively
  The degree of patient satisfaction was assessed on a 5-point Likert scale (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of adverse events | at 8 weeks postoperative and 12 weeks postoperative
  Incidence of adverse events such as bradycardia, hypotension, postoperative nausea and vomiting (PONV) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed s abdelgalil, MD, Principal Investigator — assistant professor
Locations (1):
- National cancer institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.